CLINICAL TRIAL: NCT03035097
Title: Deployment-Related Lung Disease Research Database and Biorepository
Status: Recruiting | Type: Observational
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Cecile Rose Professor of Medicine, Principal Investigator, National Jewish Health
Other Study IDs: HS-2689
Record Dates: First submitted 2017-01-04; First posted 2017-01-27 (Estimated); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis | interventions — Biological Specimen Banks

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — If patients consent to having blood and tissue collected for the biorepository, the samples will be collected during a clinic visit. Two DNA PAXgene tubes will be used to collect 17ml of blood and two RNA PAXgene tubes would be used to collect 5 ml of blood. In addition, excess bronchoalveolar lavage (BAL) fluid from a clinically-indicated bronchoscopy would also be collected. Blood and BAL fluid will be frozen and stored in -80 degree C freezers in the Occupational Medicine Laboratory until processed. If a patient will have a surgical or transbronchial biopsy as part of his or her clinical evaluation, any excess lung tissue that has been formalin-fixed and paraffin-embedded will also be collected and stored in the Occupational Medicine facilities.
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Other: Biorepository — One-time blood draw for blood to be stored in a biorepositoy

SUMMARY:
The purpose of this research study is to establish a research database and biorepository for patients at National Jewish Health (NJH) who served in Operation Iraqi Freedom (OIF) or Operation Enduring Freedom (OEF). This study will also include civilian contractors who worked as part of these military operations in Iraq or Afghanistan. The biorepository would store blood samples obtained from these patients during a clinic visit. The research database would store prospectively and retrospectively collected clinical and exposure data that would enable us to comprehensively characterize each case.

DETAILED DESCRIPTION:
If informed consent is obtained, test results and other information collected for clinical reasons will be entered in a research database designed and maintained by DEOHS staff. The clinical data collected are part of the routine diagnosis and care of these patients. No additional procedures are required for the purpose of this research database. Collection of symptom and exposure data using a questionnaire designed for this study.

All NJH patients who served in southwest Asia will be approached for inclusion in the study. This will also attempt to contact patients evaluated previously at NJH for deployment-related lung disease to obtain informed consent to include data from their medical record and the research questionnaire in the database.

ELIGIBILITY:
Inclusion Criteria:

* Served in the southwest Asia wars

Exclusion Criteria:

* Did not served in the southwest Asia wars

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who served in the southwest Asia will be approached for inclusion in the study. If patients agree to participate in the biorepository, a one-time blood draw will occur. If the subject has had a previous bronchoscopy or a surgical lung biopsy and has excess samples the study would collect those to add to the biorepository.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-02; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
collect symptom and exposure data | Up to 24 months
  each subject will complete a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zell-Baran LM, Meehan R, Wolff J, Strand M, Krefft SD, Gottschall EB, Macedonia TV, Gross JE, Sanders OL, Pepper GC, Rose CS. Military Occupational Specialty Codes: Utility in Predicting Inhalation Exposures in Post-9/11 Deployers. J Occup Environ Med. 2019 Dec;61(12):1036-1040. doi: 10.1097/JOM.0000000000001731. PMID 31592941
- [Background] Krefft SD, Wolff J, Zell-Baran L, Strand M, Gottschall EB, Meehan R, Rose CS. Respiratory Diseases in Post-9/11 Military Personnel Following Southwest Asia Deployment. J Occup Environ Med. 2020 May;62(5):337-343. doi: 10.1097/JOM.0000000000001817. PMID 31977922